CLINICAL TRIAL: NCT05196165
Title: Clinical Survey Study to Assess Physical Function and the Incidence of Hypoglycemia in Patients 1 Year of Age and Over With GSD III
Brief Title: Clinical Survey Study to Assess Physical Function and the Incidence of Hypoglycemia in Participants With Glycogen Storage Disease Type III
Status: Terminated | Type: Observational
Why Stopped: Sponsor decision not related to safety concerns
Sponsor: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: UX053-CL002
Record Dates: First submitted 2021-12-10; First posted 2022-01-19 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Glycogen Storage Disease Type III
MeSH Terms: conditions — Glycogen Storage Disease Type III

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No Intervention — No investigational product (IP) will be administered in this study

SUMMARY:
The primary objective of this study is to evaluate the incidence of hypoglycemia in adult and pediatric participants with glycogen storage disease type III (GSD III).

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of GSD III, confirmed by amylo-alpha-1,6-glucosidase 4-alpha-glucanotransferase (AGL) sequencing or glycogen debranching enzyme (GDE) enzymatic testing

Key Exclusion Criteria:

* Participant is unwilling to remain blinded to continuous glucose monitor (CGM) data for the first 13 weeks of the study, or the Investigator determines that blinding would compromise subject safety
* Presence or history of any condition that, in the view of the Investigator, would interfere with participation or pose undue risk
* Use of any IP or investigational medical device within 30 days or 5.5 half-lives, whichever is longer, prior to screening, or during the study

Note: Other criteria may apply per protocol

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study aims to enroll at least 5 participants from each of the following age groups: 1-5 years, 6-12 years, 12-17 years, and ≥ 18 years.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2022-05-20 (Actual); Primary Completion 2023-03-02 (Actual); Study Completion 2023-03-02 (Actual)

PRIMARY OUTCOMES:
Number of Hypoglycemic Events During the 26-week Observation Period | Week 26

SECONDARY OUTCOMES:
Bayley Scales of Infant and Toddler Development (Bayley-4) Fine Motor and Gross Motor Domain Scores | Up to Week 26
Bruininks-Oseretsky Test of Motor Proficiency (BOT-2) Strength and Agility Scores | Up to Week 26
Number of Times the Participant can Rise from a Seated to a Standing Position in a 30-second Period, as Measured by the Site-to-Stand (STS) Test | Up to Week 26
Percent Predicted Muscle Strength as Measured by Handheld Dynamometry (HHD) | Up to Week 26
Ankle Dorsiflexion, Measured Bilaterally Using Goniometry | Up to Week 26
Percent Predicted Distance Walked as Measured by 6-minute Walk Test (6MWT) and 12-minute Walk Test (12MWT) | Up to Week 26
GNE Myopathy Functional Activities Scale (GNEM-FAS) Expanded Version Domain Scores and Total Score | Up to Week 26

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Ultragenyx Pharmaceutical Inc
Locations (4):
- United States (3):
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - University of Texas, Houston, Texas
- University of Groningen Beatrix Children's Hospital, Groningen, Netherlands

REFERENCES:
- See also: Patient Advocacy at Ultragenyx: Glycogen Storage Disease Type III (GSDIII) — https://ultrarareadvocacy.com/conditions-we-study/glycogen-storage-disease-type-iii-gsdiii/